CLINICAL TRIAL: NCT07339553
Title: A Phase II Clinical Study of Zeprumetostat Combined With Fuzuloparib in the Treatment of Patients With Advanced or Recurrent Ovarian Epithelial Carcinoma
Brief Title: Clinical Study of EZH2 Inhibitor Combined With PARP Inhibitor in the Treatment of Patients With Advanced or Recurrent Epithelial Ovarian Cancer.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Hongyan Guo, Director, Gynecologic Oncology Department; Chief Physician, Peking University Third Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M20250852
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Ovariancancer; Platinum-sensitive Recurrent
Keywords: EZH2 Inhibitor; PARP Inhibitor; SHR2554; Zeprumetostat Tablets; Platinum-sensitive recurrent ovarian cancer
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Phase 1: Fuzuloparib Monotherapy Dose: 150 mg, twice daily (bid), orally (po). Duration: Administration for 2 to 4 weeks, until hematological toxicity recovers to pre-enrollment criteria, after which Phase 2 combination therapy may commence.
  Phase 2: Zeprumetostat Tablets in Combination with Fuzuloparib Dose: Zeprumetostat Tablets 250 mg, bid, po, Fuzuloparib 100 mg, bid, po. Duration: Treatment continues until disease progression, unacceptable toxicity, or other protocol-specified reasons for treatment discontinuation occur.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Phase 1: Fuzuloparib Monotherapy Dose: 150 mg, twice daily (bid), orally (po). Duration: Administration for 2 to 4 weeks, until hematological toxicity recovers to pre-enrollment criteria, after which Phase 2 combination therapy may commence.
  Phase 2: Zeprumetostat Tablets in Combination with Fuzuloparib Dose: Zeprumetostat Tablets 250 mg, bid, po, Fuzuloparib 100 mg, bid, po. Duration: Treatment continues until disease progression, unacceptable toxicity, or other protocol-specified reasons for treatment discontinuation occur.
  Interventions: Drug: Treatment

INTERVENTIONS:
Drug: Treatment — Phase 1: Fuzuloparib Monotherapy Dose: 150 mg, twice daily (bid), orally (po). Duration: Administration for 2 to 4 weeks, until hematological toxicity recovers to pre-enrollment criteria, after which Phase 2 combination therapy may commence.
  Phase 2: Zeprumetostat Tablets in Combination with Fuzuloparib Dose: Zeprumetostat Tablets 250 mg, bid, po, Fuzuloparib 100 mg, bid, po. Duration: Treatment continues until disease progression, unacceptable toxicity, or other protocol-specified reasons for treatment discontinuation occur.

SUMMARY:
This study evaluates the efficacy and safety of Zeprumetostat in combination with Fuzuloparib for the treatment of patients with advanced or recurrent ovarian epithelial carcinoma, with the primary endpoint being Objective Response Rate (ORR).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years.
* Histologically or cytologically confirmed ovarian carcinoma with FIGO Stage III-IV disease, or recurrent ovarian epithelial carcinoma (any stage or timing of recurrence), with genetic testing results indicating BRCA1/2 wild-type.
* At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors version 1.1 (computed tomography scan showing the longest diameter of a non-lymph node tumor lesion is no less than 10 millimeters, or the short axis of a lymph node lesion is no less than 15 millimeters), or abnormal cancer antigen 125 levels, or presence of ascites, as confirmed by the investigator.
* Eastern Cooperative Oncology Group (ECOG) Performance Status score between 0 and 2; expected survival of at least 3 months.
* Adequate function of major organs, with screening laboratory test results meeting the following requirements:

Complete Blood Count criteria must be met:

A. Hemoglobin ≥ 80 grams per liter; B. Absolute neutrophil count ≥ 1.5 × 10⁹ per liter; C. Platelet count ≥ 80 × 10⁹ per liter.

Biochemistry criteria must meet the following standards:

A. Total bilirubin < 1.5 times the upper limit of normal; B. Alanine aminotransferase and aspartate aminotransferase < 2.5 times the upper limit of normal, and < 5 times the upper limit of normal for patients with liver metastases; C. Serum creatinine ≤ 1.5 times the upper limit of normal or endogenous creatinine clearance > 60 milliliters per minute (calculated by the Cockcroft-Gault formula); D. Urine protein < 2+ or 24-hour urinary protein quantification < 1 gram.

* Signed written informed consent, with anticipated good compliance to the study protocol.
* After completion of the first phase (Fuzuloparib monotherapy), subjects who experience hematological toxicity may proceed to the second phase (combination therapy) only after the investigator determines that the hematological toxicity has recovered to meet the enrollment criteria.

Exclusion Criteria:

* Patients with active brain metastases.
* Use of immunosuppressive drugs within the 28 days prior to enrollment, excluding intranasal and inhaled corticosteroids or physiological doses of systemic corticosteroids (i.e., no more than 10 mg/day of prednisolone or equivalent doses of other corticosteroids for physiological replacement).
* Systemic treatment with Chinese herbal medicines with approved anti-tumor indications or drugs with immunomodulatory effects (including thymosin, interferon, interleukin; except for local use in controlling pleural effusion) within 2 weeks prior to the first dose.
* History of severe cardiovascular diseases: myocardial ischemia of grade II or higher or myocardial infarction, poorly controlled arrhythmias (including corrected QT interval ≥ 470 ms in females); cardiac dysfunction of grade III to IV according to the New York Heart Association classification (see Appendix 3), or left ventricular ejection fraction less than 50% as indicated by cardiac ultrasound.
* Concurrent severe infection within 4 weeks prior to the first dose, or unexplained fever > 38.5°C during screening/prior to the first dose; or major surgical procedure within 3 weeks prior to the first dose.
* Presence of active autoimmune disease or immunodeficiency, including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, rheumatoid arthritis, inflammatory bowel disease, hypophysitis, vasculitis, nephritis, etc.
* Subjects requiring systemic therapy such as bronchodilators with suboptimal asthma control.
* Subjects who have undergone or plan to undergo solid organ or hematopoietic system transplantation during the study period (except for corneal transplantation).
* Current participation in an interventional clinical study, or treatment with other investigational drugs or devices within 4 weeks prior to the first dose; or not having fully recovered from toxicities and/or complications caused by any previous intervention prior to the first dose.
* Uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 110 mmHg despite optimal medical therapy).
* Abnormal coagulation function (international normalized ratio > 1.5, or prothrombin time > upper limit of normal + 4 seconds, or activated partial thromboplastin time > 1.5 times the upper limit of normal), bleeding tendency, or current use of thrombolytic or anticoagulant therapy.
* History of psychoactive drug abuse and inability to abstain, or history of mental disorders.
* History of hereditary or acquired bleeding disorders or coagulation dysfunction (subject to investigator's judgment on eligibility).
* Concomitant use of strong cytochrome P450 3A4 inhibitors (e.g., itraconazole, telithromycin, clarithromycin, etc.), moderate cytochrome P450 3A4 inhibitors (e.g., ciprofloxacin, erythromycin, fluconazole, etc.), strong cytochrome P450 3A4 inducers (e.g., phenobarbital, enzalutamide, phenytoin, rifampin, etc.), or moderate cytochrome P450 3A4 inducers (e.g., bosentan, modafinil, etc.). Required washout period prior to initiation of study treatment is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
* Prior exposure to other enhancer of zeste homolog 2 inhibitors.
* History of cerebrovascular accident or transient ischemic attack within the past 6 months.
* Any other condition that, in the judgment of the investigator, increases the risk associated with study participation or administration of the investigational product, and would make the patient unsuitable for inclusion in the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2026-01-04 (Estimated); Primary Completion 2029-01-30 (Estimated); Study Completion 2029-02-26 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 12 months
  The proportion of patients achieving tumour volume reduction meeting predetermined criteria (RECIST 1.1) and maintaining this reduction for a specified duration (typically at least four weeks), encompassing both complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
Progression-Free Survival | 24 months
  The time from the start of treatment to tumour progression or death from any cause, whichever occurs first.
Overall Survival | 36 months
  The time from the commencement of treatment to death from any cause.

IPD SHARING:
Plan to Share IPD: No